CLINICAL TRIAL: NCT04248348
Title: Metaxa's Thromboprophylaxis Program in Oncological & Surgical Patients
Brief Title: Metaxa Hospital THromboprophylaxis Program in Oncological & Surgical Patients
Acronym: MeTHOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Metaxa Hospital (Other)
Responsible Party: Principal Investigator, Nikolaos Ziras, Head of Oncology Clinic, Metaxa Hospital
Other Study IDs: 2394-05/02/2019
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Thrombosis; Solid Cancer
Keywords: Thrombosis; Cancer; Heparin, Low Molecular Weight
MeSH Terms: conditions — Thrombosis; Neoplasms | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Low Molecular Weight Heparin — Cancer patients will be protected against thrombosis using Low Molecular Weight Heparin (LMWH)

SUMMARY:
During MeTHOS study will be collected Real World Data the clinical practice regarding Thromboprophylaxis in high thrombotic risk solid tumors patients undergoing surgical and /or chemotherapeutical treatment, for one year following the protocol initiation date.

Specifically focus will be on the following:

* Number of thrombotic events
* Anti-thrombotic management dosage & duration
* Any bleedings related to anticoagulation
* Patients' adherence and compliance

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic and genitourinary) undergoing surgery
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Life expectancy >6 months
5. Signed informed consent

Exclusion Criteria

1. Patients who were not diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic and genitourinary) undergoing surgery
2. Age < 18 years
3. ECOG performance status >2
4. Life expectancy <6 months
5. Not signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of thrombotic events | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Measure the number of thrombotic events in the population
Number of bleedings related to anticoagulation | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Measure the number of observed bleeding events caused by the anticoagulation treatment

SECONDARY OUTCOMES:
Anticoagulation drug dosage | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Record the antithrombotic drug dosage (IU/day), aiming to investigate the role of dosage for thrombotic events and bleedings (primary outcomes)
Anticoagulation drug duration | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Record the antithrombotic drug duration (in days). The aim is to investigate the role of antithrombotic duration for thrombotic events and bleedings (primary outcomes)
Patients' compliance to anticoagulation treatment | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Record the compliance of patients' in antithrombotic treatment. A patient is considered to be compliant if the anticoagulation treatment was administered as prescribed (usually every day), otherwise it is non-compliant. The aim is to investigate the role of patient compliance for thrombotic events and bleedings (primary outcomes).
Anticoagulation drug agent | Each subject's participation will last from inclusion (enrolment visit) to follow up visit (if applicable; four weeks post hospital discharge)
  Record the anticoagulation drug agent. The aim is to investigate the role of different agents for thrombotic events and bleedings (primary outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Ziras, MD, Study Chair — Metaxa Hospital; Spyridon Xynogalos, MD, Principal Investigator — Metaxa Hospital
Locations (1):
- Metaxa Hopital, Piraeus, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Data may be provided upon a reasonable request.

REFERENCES:
- [Derived] Xynogalos S, Simeonidis D, Papageorgiou G, Pouliakis A, Charalambakis N, Lianos E, Mazlimoglou E, Liatsos AN, Kosmas C, Ziras N. Can thromboprophylaxis build a link for cancer patients undergoing surgical and/or chemotherapy treatment? The MeTHOS cohort study. Support Care Cancer. 2022 Aug;30(8):6973-6984. doi: 10.1007/s00520-022-07096-1. Epub 2022 May 12. PMID 35552827

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04248348/Prot_SAP_000.pdf